CLINICAL TRIAL: NCT01100684
Title: A 12-Week, Randomized, Double-Blind, Placebo-Controlled Study of Asimadoline in Subjects With Diarrhea-Predominant Irritable Bowel Syndrome (D-IBS)
Brief Title: Study of Asimadoline to Treat Diarrhea-Predominant Irritable Bowel Syndrome (D-IBS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tioga Pharmaceuticals (Industry)
Collaborators: RTI Health Solutions (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASMP3001
Record Dates: First submitted 2010-04-06; First posted 2010-04-09 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Diarrhea Predominant Irritable Bowel Syndrome
Keywords: diarrhea predominant irritable bowel syndrome
MeSH Terms: interventions — asimadoline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): 0.5 mg asimadoline bid
  Interventions: Drug: Asimadoline
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Asimadoline — 0.5 mg Asimadoline BID
  Other Names: EMD 61 753; EMR 63 320
  Arms: Treatment
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether asimadoline is safe and effective at treating D-IBS.

DETAILED DESCRIPTION:
The primary objective of the study is to compare the efficacy of the two treatments with respect to improvement in IBS-related abdominal pain severity and reduction in stool frequency. During the 12-week treatment period, daily IBS-related abdominal pain severity score and daily frequency of bowel movements will be averaged over each week to determine average values for each endpoint. For each subject, weekly response to treatment will be based on the following parameters:

* Decrease from baseline of at least 30% in the average IBS-related daily abdominal pain severity score
* Decrease from baseline of at least 25% in the average number of daily bowel movements A subject must meet both criteria to be considered a weekly responder. The primary efficacy endpoint is based on an "overall study responder," defined as a subject having 6 or more weeks of weekly response to treatment out of the 12 weeks in the treatment period. Overall study responder will be stratified by timing of bowel preparation and endoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Signs and dates a written informed consent form.
2. Male and female subjects aged 18-79 who are fluent in English
3. All subjects must use protocol specified contraceptive measures
4. The subject is or has been diagnosed with IBS with symptom onset at least 6 months prior to diagnosis. IBS is defined as the subject having recurrent abdominal pain or discomfort at least 3 days per month in the past 3 months associated with at least two of the following symptoms:

   Improvement with defecation Onset associated with a change in frequency of stool Onset associated with a change in form (appearance) of stool
5. The subject has been diagnosed with diarrhea-predominant IBS
6. Within 2 years of the randomization visit, the subject has normal results from a flexible sigmoidoscopy, a colonoscopy, or a barium enema plus flexible sigmoidoscopy, according to the subject's age by a specified algorithm.

Exclusion Criteria:

1. The subject exhibits evidence of a biochemical or structural abnormality of the digestive tract.
2. Subject has a concurrent illness or disability (excluding IBS) that may affect the interpretation of clinical efficacy and/or safety data or otherwise contraindicates participation in this clinical study (e.g., an unstable cardiovascular, renal, hepatic, pulmonary, endocrine, metabolic, GI, hematological, or neurological condition).
3. The subject has a family history of prolonged QT syndrome.
4. The subject has been diagnosed with a major psychiatric disorder.
5. The subject has a history of alcohol or substance abuse within the past 2 years.
6. The subject has a history or current evidence of laxative abuse
7. The subject has a positive stool sample for ova or parasite.
8. The subject has used an investigational drug or participated in an investigational study within 30 days of screening.
9. The subject refuses to discontinue one (or more) prohibited medications at least 7 days prior to the screening visit.
10. The subject refuses to maintain a stable dose of one (or more) allowable concurrent medications for at least 30 days prior to the screening visit.
11. The subject is a pregnant woman or a woman who is breast feeding.
12. The subject is unable or unwilling to follow directions or use the electronic diary system.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 611 (Actual)
Dates: Start 2010-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
12 Week Abdominal Pain and Stool (APS) Frequency Responder | Weekly responder based on patient assessments made daily in each week of the 12-week Treatment Period to determine 12 week APS responder
  A study responder is a subject who has both a decrease from baseline of IBS-related abdominal pain and a decrease from baseline of daily bowel movements

SECONDARY OUTCOMES:
Compare the two treatment groups with respect to IBS-related abdominal pain | Up to 12 weeks
Compare the two treatment groups with respect to stool frequency | Up to 12 weeks
Compare the two treatment groups with respect to stool urgency | Up to 12 weeks
Compare the two treatment groups with respect to IBS symptoms | up to 12 weeks
Compare the two treatment groups with respect to stool consistency scores | Up to 12 weeks
  Using the Bristol Stool Form Scale
Incidence of adverse events as a measure of tolerability | Up to 16 weeks
Abnormalities of laboratory tests as a measure of tolerability | Up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Allen Mangel, M.D.Ph.D., Study Chair — CMO
Locations (142):
- United States (142):
  - North Alabama Research Center, LLC, Athens, Alabama
  - Alliance Clinical Research, Birmingham, Alabama
  - Medical Affliated Research Center, Inc., Huntsville, Alabama
  - Saadat Ansari MD LLC, Huntsville, Alabama
  - Connect Clinical Research Center, Chandler, Arizona
  - Digestive Health Research Unit, Scottsdale, Arizona
  - Adobe Clinical Research, LLC, Tucson, Arizona
  - ACRC/Arizona Clinical Research Center, Inc., Tucson, Arizona
  - Genova Clinical Research, Tucson, Arizona
  - W/C Clinical Research, Tucson, Arizona
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Arkansas Gastroenterology, Sherwood, Arkansas
  - Providence Clinical Research, Burbank, California
  - GW Research Inc,, Chula Vista, California
  - La Jolla Clinical Research, Inc, Chula Vista, California
  - Discovery Clinical Research, Encinitas, California
  - Digestive & Liver Disease Specialist, Garden Grove, California
  - Collaborative Neuroscience Network Inc, Long Beach, California
  - California Gastroenterology Associates, Madera, California
  - Community Clinical Trials, Orange, California
  - Sutter Medical Group Gastroenterology, Sacramento, California
  - Medical Center for Clinical Research, San Diego, California
  - Medical Associates Research Group, Inc., San Diego, California
  - Westlake Medical Research, Westlake Village, California
  - Lynne Institute of the Rockies, Colorado Springs, Colorado
  - Arapahoe Gastroenterology, Littleton, Colorado
  - Lynn Institute of Pueblo, Pueblo, Colorado
  - Rocky Mountain Gastroenterology Associates, Thornton, Colorado
  - Danbury Clinical Research, LLC, Danbury, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Consultants for Clinical Research of South Florida, Boynton Beach, Florida
  - Meridien Research, Brookville, Florida
  - BioPharma Research, Coral Gables, Florida
  - Riverside Clinical Research, Edgewater, Florida
  - A.G.A. Clinical Trials, Hialeah, Florida
  - Altus Research, Lake Worth, Florida
  - Center for Advanced Gastroenterology, Maitland, Florida
  - FIRC, Miami, Florida
  - DMI Research, Pinellas Park, Florida
  - Accord Clinical Research, LLC, Port Orange, Florida
  - International Clinical Research-US,LLC, Sanford, Florida
  - Lakeview Medical Research, Summerfield, Florida
  - Venra Clinical Studies, LLC, Wellington, Florida
  - Alliance Clinical Research, Winter Park, Florida
  - Atlanta Center for Gastroenterology, Decatur, Georgia
  - Tri County Research, Hartwell, Georgia
  - Northwest Gastroenterologist S.C., Arlington Heights, Illinois
  - Illinois Center for Clinical Research, Chicago, Illinois
  - Southwest Gastroenterology, Oak Lawn, Illinois
  - Elkhart Clinic, LLC/Indiana Medical Research, LLC, Elkhart, Indiana
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Mercy Gastroenterology Clinic, Clive, Iowa
  - Gastrointestinal Clinic of Quad Cities, Davenport, Iowa
  - Heartland Research Associates, LLC, Newton, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Graves-Gilbert Clinic, Bowling Green, Kentucky
  - Tri-State Gastroenterology Associates, PSC, Crestview Hills, Kentucky
  - Hometown Urgent Care and Research, Hebron, Kentucky
  - The Research Group of Lexington, LLC, Lexington, Kentucky
  - University of Louisville Medical-Dental Complex, Louisville, Kentucky
  - Tover Health Systems Center for Clinical Research, Madisonville, Kentucky
  - Investigative Clinical Research, Annapolis, Maryland
  - Meritus Center for Clinical Resarch, Hagerstown, Maryland
  - Spectrum Clinical Research Inc., Towson, Maryland
  - Commonwealth Clinical Studies, Brockton, Massachusetts
  - NECCR Internal Medicine and Cardiology Associates LLC, Fall River, Massachusetts
  - ActivMed Practices and Research, Haverhill, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Saginaw Valley Medical Research Group, LLC, Saginaw, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Gastrointestinal Accociates, PA, Jackson, Mississippi
  - Digestive Research Specialist, Tupelo, Mississippi
  - Midwest Center for Clinical Research, Lees Summit, Missouri
  - Center for Digestive and Liver Diseases, Inc., Mexico, Missouri
  - St. Louis Center for Clinical Research, St Louis, Missouri
  - Montana Health Research Institute, Inc., Billings, Montana
  - Dr. Meera Dewan PC, Omaha, Nebraska
  - Anderson & Collins Clinical Research, Edison, New Jersey
  - South Jersey Gastroenterology. P.A., Marlton, New Jersey
  - Atlantic Research Affiliates, Morristown, New Jersey
  - Life Medi-Research, Brooklyn, New York
  - Long Island Clinical Research Associates, LLP, Great Neck, New York
  - Long Island Gastrointestinal Research Group, Great Neck, New York
  - Winthrop University Hospital Clinical Trials Center, Mineola, New York
  - Research Associates of New York, New York, New York
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - Gastrointestinal Research Associates, LLC, Setauket, New York
  - The UNC Center for Functional GI and Motility Disorders, Chapel Hill, North Carolina
  - PMG Research of Charlotte, LLC, Charlotte, North Carolina
  - LeBauer Research Associates, P.A., Greensboro, North Carolina
  - PMG Research of Hickory, LLC, Hickory, North Carolina
  - Peters Medical Research, High Point, North Carolina
  - Kinston Medical Specialist, P.A., Kinston, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Trial Management Associates LLC, Wilmington, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Akron Gastroenterology Associates, Akron, Ohio
  - Gastroenterology Research Consultants of Greater Cincinnati, Cincinnati, Ohio
  - Hometown Urgent Care, Columbus, Ohio
  - Hometown Urgent Care, Dayton, Ohio
  - Hometown Urgent Care and Research, Groveport, Ohio
  - Hometown Urgent Care and Research, Miamisburg, Ohio
  - Physicians Research, Inc, Zanesville, Ohio
  - Journey Clinical Research, Duncan, Oklahoma
  - Central Sooner Research, Norman, Oklahoma
  - Oklahoma Foundation for Digestive Research, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Northwest Gastroenterology Clinic, LLC, Portland, Oregon
  - Safe Harbor Clinical Research, East Providence, Rhode Island
  - Southeast Medical Research, Charleston, South Carolina
  - SC Clinical Research, LLC, Columbia, South Carolina
  - Coastal Carolina Research Center in Goose Creek, Goose Creek, South Carolina
  - Hillcrest Clinical Research, LLC, Simpsonville, South Carolina
  - Midwest Medical Care, Sioux Falls, South Dakota
  - Gastroenterology Associates, Bristol, Tennessee
  - ClinSearch, LLC, Chattanooga, Tennessee
  - Alpha Clinical Research, Clarksville, Tennessee
  - Memphis Gastroenterology Group, Germantown, Tennessee
  - Associates in Gastroenterology, Hermitage, Tennessee
  - Gastroenterology Associates Clinical Research, Kingsport, Tennessee
  - Columbia Medical Group -The First Clinic, Inc., Nashville, Tennessee
  - Dial Research Associates, INC, Nashville, Tennessee
  - TN Medical Research, Spring Hill, Tennessee
  - Research Across America/ Family Medicine Associates of Texas, Carrollton, Texas
  - Corsicana Medical Research, PLLC, Corsicana, Texas
  - Texas University Health Sciences Center, El Paso, Texas
  - Gastroenterology Consultants, P.A., Houston, Texas
  - Houston S. Endoscopy and Research Center, Houston, Texas
  - Pioneer Research Solutions, Inc, Houston, Texas
  - Digestive Health Associates of Texas, Plano, Texas
  - Sun Research Institute, San Antonio, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Advanced Research Institute, Clinton, Utah
  - Advanced Research Institute, Logan, Utah
  - Advanced Research Institute, Ogden, Utah
  - Advanced Research Institute, Sandy City, Utah
  - Gastroenterology, Ltd., Virginia Beach, Virginia
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin